CLINICAL TRIAL: NCT05991453
Title: Trajectories of Recovery After Intravenous Propofol Versus Inhaled VolatilE Anesthesia Trial
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202304082
Record Dates: First submitted 2023-06-23; First posted 2023-08-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Surgery-Complications; Anesthesia Complication; Anesthesia Awareness; Anesthesia; Surgery; Quality of Life; Pain, Postoperative; Anesthesia Morbidity
MeSH Terms: conditions — Intraoperative Awareness; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol total intravenous anesthesia (TIVA) (Active Comparator): No administration of inhaled agent.
  Interventions: Other: Anesthetic technique Propofol TIVA
- inhaled volatile general anesthesia (INVA) (Active Comparator): Must administer inhaled agent.
  Interventions: Other: Anesthetic technique inhaled agent

INTERVENTIONS:
Other: Anesthetic technique Propofol TIVA — Propofol TIVA no inhaled agent
  Other Names: Propofol TIVA
  Arms: Propofol total intravenous anesthesia (TIVA)
Other: Anesthetic technique inhaled agent — Must administer inhaled agent.
  Other Names: Inhaled agent
  Arms: inhaled volatile general anesthesia (INVA)

SUMMARY:
The investigators will conduct a 13,000-patient randomized multi-center trial to determine (i) which general anesthesia technique yields superior patient recovery experiences in any of three surgical categories ((a) major inpatient surgery, (b) minor inpatient surgery, (c) outpatient surgery) and (ii) whether TIVA confers no more than a small (0.2 %) increased risk of intraoperative awareness than INVA in patients undergoing both outpatient and inpatient surgeries

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following criteria:

1. Aged 18 years or older
2. Undergoing elective non-cardiac surgery expected to last ≥ 60 min requiring general anesthesia with a tracheal tube or laryngeal mask airway (or similar supra-glottic device)

Exclusion Criteria

Patients will not be enrolled if any of the following criteria are met:

1. Inability to provide informed consent in English (at all study sites) or Spanish (at sites where Spanish consent is provided as an option)
2. Pregnancy (based on patient report or positive test on the day of surgery)
3. Surgical procedure requiring general, regional, neuraxial anesthesia administered by an anesthesia clinician (anesthesiologist, CRNA, anesthesiology assistant) occurring within 30 days prior to or planned to occur within 30 days after surgery date
4. Contraindication to propofol TIVA or INVA (for example, documented allergy to propofol, history of severe postoperative nausea or vomiting, concern for or history of malignant hyperthermia) based on self-report
5. Surgical procedures requiring a specific general anesthesia technique (for example, TIVA required for neuromonitoring).
6. Locally approved, written protocol mandating a particular anesthetic technique
7. History of possible or definite intraoperative awareness during general anesthesia based on patient self-report
8. Planned postoperative intubation
9. Current incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13000 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 1 after major inpatient surgery | Postoperative day 1
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 1 after minor inpatient surgery | Postoperative day 1
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 1 after outpatient surgery | Postoperative day 1
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Incidence of definite intraoperative awareness with recall | Postoperative day 30
  The modified Brice questionnaire is used to screen for intraoperative awareness. A positive screen (a patient who reports remembering anything between going to sleep for their surgical procedure and waking up after) on the modified Brice questionnaire is followed by a structured interview. A panel of expert adjudicators determines whether or not this was definite intraoperative awareness.

SECONDARY OUTCOMES:
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 0 after major inpatient surgery | postoperative day 0
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 0 after minor inpatient surgery | postoperative day 0
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 0 after outpatient surgery | postoperative day 0
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 2 after major inpatient surgery | postoperative day 2
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 2 after minor inpatient surgery | postoperative day 2
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 2 after outpatient surgery | postoperative day 2
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 7 after major inpatient surgery | postoperative day 7
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 7 after minor inpatient surgery | postoperative day 7
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Patient Reported Quality of Recovery-15 (QOR15) score on postoperative day 7 after outpatient surgery | postoperative day 7
  The QOR15 instrument measures quality of recovery with a score of 0 - 150 points where the higher the score the better quality of recovery.
Days Alive and at Home at 30 days after major inpatient surgery | postoperative day 30
  Patient hospital length of stay after the surgery is documented. A patient completed survey assesses hospital re-admission since discharge from surgery and days spent in the hospital since original discharge.
Days Alive and at Home at 30 days after minor inpatient surgery | postoperative day 30
  Patient hospital length of stay after the surgery is documented. A patient completed survey assesses hospital re-admission since discharge from surgery and days spent in the hospital since original discharge.
Days Alive and at Home at 30 days after outpatient surgery | postoperative day 30
  Patient hospital length of stay after the surgery is documented. A patient completed survey assesses hospital re-admission since discharge from surgery and days spent in the hospital since original discharge.
Incidence of delirium on postoperative day 0 after major inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium.
Incidence of delirium on postoperative day 0 after minor inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium.
Incidence of delirium on postoperative day 0 after outpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium.
Incidence of delirium on postoperative day 1 after major inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium.
Incidence of delirium on postoperative day 1 after minor inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium.
Delirium Severity Score on postoperative day 0 after major inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The 3D-CAM severity score is calculated by adding 1 point for each positive item noted in questions 1-20. The score is calculated out of 20 points - a higher score indicates a higher severity.
Delirium Severity Score on postoperative day 0 after minor inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The 3D-CAM severity score is calculated by adding 1 point for each positive item noted in questions 1-20. The score is calculated out of 20 points - a higher score indicates a higher severity.
Delirium Severity Score on postoperative day 0 after outpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The 3D-CAM severity score is calculated by adding 1 point for each positive item noted in questions 1-20. The score is calculated out of 20 points - a higher score indicates a higher severity.
Delirium Severity Score on postoperative day 1 after major inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The 3D-CAM severity score is calculated by adding 1 point for each positive item noted in questions 1-20. The score is calculated out of 20 points - a higher score indicates a higher severity.
Delirium Severity Score on postoperative day 1 after minor inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The 3D-CAM severity score is calculated by adding 1 point for each positive item noted in questions 1-20. The score is calculated out of 20 points - a higher score indicates a higher severity.
Incidence of Subsyndromal delirium on postoperative day 0 after major inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The presence of at least 1 feature is indicative of subsyndromal delirium.
Incidence of Subsyndromal delirium on postoperative day 0 after minor inpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The presence of at least 1 feature is indicative of subsyndromal delirium.
Incidence of Subsyndromal delirium on postoperative day 0 after outpatient surgery | postoperative day 0
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The presence of at least 1 feature is indicative of subsyndromal delirium.
Incidence of Subsyndromal delirium on postoperative day 1 after major inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The presence of at least 1 feature is indicative of subsyndromal delirium.
Incidence of Subsyndromal delirium on postoperative day 1 after minor inpatient surgery | postoperative day 1
  The 3D Confusion Assessment Method (3DCAM) assesses four key features of delirium. The presence of at least 1 feature is indicative of subsyndromal delirium.
Health-related quality-of-life on postoperative day 30 after major inpatient surgery | postoperative day 30
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 30 after minor inpatient surgery | postoperative day 30
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 30 after outpatient surgery | postoperative day 30
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 90 after major inpatient surgery | postoperative day 90
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 90 after minor inpatient surgery | postoperative 90 days
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 90 after outpatient surgery | postoperative day 90
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 180 after major inpatient surgery | postoperative day 180
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 180 after minor inpatient surgery | postoperative day 180
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 180 after outpatient surgery | postoperative day 180
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 365 after major inpatient surgery | postoperative day 365
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 365 after minor inpatient surgery | postoperative day 365
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Health-related quality-of-life on postoperative day 365 after outpatient surgery | postoperative day 365
  EQ-5D-5L will be used as a measure of health-related quality-of-life. For scoring guidelines please see the manual https://euroqol.org/wp-content/uploads/2023/03/EQ-5D-5LUserguide-08-0421.pdf
Functional status on postoperative day 30 after major inpatient surgery. | postoperative day 30
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Functional status on postoperative day 30, after minor inpatient surgery. | postoperative day 30
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Functional status on postoperative day 30, after outpatient surgery. | postoperative day 30
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Functional status on postoperative day 90 after major inpatient surgery. | postoperative day 90
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Functional status on postoperative day 90 after minor inpatient surgery. | postoperative day 90
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Functional status on postoperative day 90 after outpatient surgery. | postoperative day 90
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a generic assessment instrument for functional status covering 6 domains of functioning: cognition, mobility, Self-care, interacting with other people, life activities, and participation.
Patient satisfaction with anesthesia on postoperative day 2 | postoperative day 2
  The Bauer questionnaire is a patient self-reported survey assessing anesthesia-related discomfort and satisfaction with anesthesia care.
Respiratory Failure on postoperative day 0 | postoperative day 0
  Respiratory failure defined as unplanned postoperative intubation or reintubation or continued mechanical ventilation > 6 hours postoperatively. Reintubation due to reoperation is excluded.
Kidney Injury on postoperative day 7 | postoperative day 7
  Kidney Injury defined as a serum creatinine increase of 50% or 0.3 mg/dl from preoperative baseline
All-Cause Mortality at POD30 | postoperative day 30
  All-Cause Mortality at POD30
All-Cause Mortality at POD90 | postoperative day 90
  All-Cause Mortality at POD90
Intraoperative Hypotension (1) | postoperative day 0
  Intraoperative Hypotension defined as cumulative duration of mean arterial pressure <55 mmHg for 20 minutes or greater.
Intraoperative Hypotension (2) | postoperative day 0
  Intraoperative hypotension defined as cumulative duration of mean arterial pressure < 65 mmHg for 20 minutes or greater.
Moderate or Severe Intraoperative Patient Movement | postoperative day 0
  Moderate or Severe Intraoperative Patient Movement is based on clinician report.
Unplanned Admission After Outpatient Surgery in an Ambulatory Setting | postoperative days 0 and 1
  Hospital admission no later than 24 hours postoperatively after outpatient surgery in a free-standing ambulatory surgery center setting
Incidence of propofol-related infusion syndrome | postoperative day 0
  Propofol related infusion syndrome, defined as acute refractory bradycardia in the presence of metabolic acidosis, and at least one of the following: rhabdomyolysis, acute kidney injury or hypertriglyceridemia, occurring after the start of propofol intraoperatively and within 6 hours postoperatively.
Incidence of malignant hyperthermia | postoperative day 0
  Malignant hyperthermia, defined as unexplained muscle rigidity, tachycardia, hypercapnia, and rapidly increasing temperature leading to metabolic acidosis, rhabdomyolysis, disseminated intravascular coagulation, and ventricular arrhythmias, occurring after the start of an inhaled volatile agent intraoperatively and within 6 hours postoperatively.

OTHER OUTCOMES:
Daily step count as measured by wearable device at baseline for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Daily step count at baseline - number of steps per day
Daily step count as measured by wearable device at baseline for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Daily step count at baseline - number of steps per day
Daily step count as measured by wearable device at baseline for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Daily step count at baseline - number of steps per day
Daily step count as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily step count as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily step count as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily step count as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily step count as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily step count as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device Daily step count: Proportion of patients within 10% of baseline, defined as steps per day
Daily standing hours as measured by wearable device at baseline for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Daily standing hours: defined as standing hours per day
Daily standing hours as measured by wearable device at baseline for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Daily standing hours: defined as standing hours per day
Daily standing hours as measured by wearable device at baseline for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Daily standing hours: defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Daily standing hours as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device.
  Daily standing hours: Proportion of patients within 10% of baseline, defined as standing hours per day
Total sleep time as measured at baseline by wearable device for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Total sleep time defined as minutes of total sleep time per day
Total sleep time as measured at baseline by wearable device for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Total sleep time defined as minutes of total sleep time per day
Total sleep time as measured at baseline by wearable device for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Total sleep time defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Total sleep time as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Total sleep time: Proportion of patients within 10% of baseline, defined as minutes of total sleep time per day
Sleep onset latency as measured by wearable device at baseline for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Sleep onset latency: defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device at baseline for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Sleep onset latency: defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device at baseline for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Sleep onset latency: defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Sleep onset latency as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Sleep onset latency: Proportion of patients within 10% of baseline, defined as minutes of sleep onset latency per day
Wake after sleep onset as measured by wearable device for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Wake after sleep onset: defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Wake after sleep onset: defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Wake after sleep onset: defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Wake after sleep onset as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Wake after sleep onset: Proportion of patients within 10% of baseline, defined as minutes of wake after sleep onset
Sleep efficiency as measured at baseline by wearable device for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Sleep efficiency: defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured at baseline by wearable device for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Sleep efficiency: defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured at baseline by wearable device for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Sleep efficiency: defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Sleep efficiency as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable
  Sleep efficiency: Proportion of patients within 10% of baseline, defined as % sleep efficiency (ranging from 0-100)
Midpoint of sleep as measured at baseline by wearable device for those scheduled for outpatient surgery. | 1 - 7 days prior to surgery
  Midpoint of sleep: defined as midpoint of sleep (time)
Midpoint of sleep as measured at baseline by wearable device for those scheduled for minor inpatient surgery. | 1 - 7 days prior to surgery
  Midpoint of sleep: defined as midpoint of sleep (time)
Midpoint of sleep as measured at baseline by wearable device for those scheduled for major inpatient surgery. | 1 - 7 days prior to surgery
  Midpoint of sleep: defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for major inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for minor inpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for outpatient surgery. | 7 - 10 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for outpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for minor inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)
Midpoint of sleep as measured by wearable device for those scheduled for major inpatient surgery. | 30 - 34 days after surgery
  Measurement of outcomes will be median values measured on their wearable device
  Midpoint of sleep: Proportion of patients within 60 minutes of baseline, defined as midpoint of sleep (time)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Kheterpal, MD, Principal Investigator — University of Michigan; Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Allison Janda, MD, Study Director — University of Michigan; Mark Neuman, MD, Study Director — University of Pennsylvania; Bethany Pennington, PharmD, Study Director — Washington University School of Medicine; Douglas Colquhoun, MBChB, Study Director — University of Michigan
Locations (20):
- United States (20):
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson, Houston, Texas
  - University of Utah - Medical, Salt Lake City, Utah
  - UVA Health, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Per the contract with the funder PCORI, the THRIVE Data Sharing Plan will be consistent with PCORI's Policy for Data Management and Data Sharing, which calls for the researchers PCORI funds to share their data sets and documentation for reanalysis and reuse. THRIVE will upload a deidentified dataset to the Patient-Centered Outcomes Data Repository (PCODR), which was created and is hosted by the Inter-University Consortium for Political and Social Research (ICPSR), a unit within the Institute for Social Research at the University of Michigan. The THRIVE study, as the Awardee, will enter into a Data Contributor Agreement (DCA) with ICPSR. The DCA governs the data deposition and establishes the Awardee's rights and obligations. The data package will be transferred to the data repository by October 1, 2028, per the contract with PCORI.
Supporting Information: Study Protocol
Time Frame: The data package will be transferred to the data repository by October 1, 2028, per the contract with PCORI.
Access Criteria: PCORI's access criteria and data sharing policy for third parties can be found here https://www.pcori.org/sites/default/files/PCORI-Policy-for-Data-Management-and-Data-Sharing.pdf
URL: https://www.pcori.org/sites/default/files/PCORI-Policy-for-Data-Management-and-Data-Sharing.pdf

REFERENCES:
- [Derived] Tellor Pennington BR, Janda AM, Colquhoun DA, Neuman MD, Kidwell KM, Spino C, Thelen-Perry S, Krambrink A, Huang S, Ignacio R, Wu Z, Swisher L, Cloyd C, Vaughn MT, Pescatore NA, Bollini ML, Mashour GA, Hassett A, Kent CD, Vlisides PE, Avidan MS, Kheterpal S; ˠTHRIVE Research Group. Trajectories of Recovery after Intravenous propofol versus inhaled VolatilE anaesthesia (THRIVE) randomised controlled trial in the USA: A protocol. BMJ Open. 2025 Sep 14;15(9):e103836. doi: 10.1136/bmjopen-2025-103836. PMID 40953862